CLINICAL TRIAL: NCT03352908
Title: Yale Swallow Protocol in Recently Extubated Patients
Brief Title: Yale Swallow Protocol in Extubated Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-1149; A539772 (Other: UW Madison); SMPH/SURGERY/SPEECH (Other: UW Madison); Protocol Version 9/28/2017 (Other: UW Madison)
Record Dates: First submitted 2017-10-30; First posted 2017-11-24 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Dysphagia
Keywords: Dysphagia; Aspiration; YSP; FEES; Swallow Problems
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- YSP: The Yale Swallow Protocol (YSP) consists of a brief cognitive screen, a brief oral motor exam, and a 3oz water challenge (subjects instructed to drink 3oz of water without stopping). Pass/fail is determined based on the subjects ability to drink the 3oz of water uninterrupted without immediate cough.
- FEES: Flexible Endoscopic Evaluation of Swallowing (FEES) uses a flexible endoscope that will be passed transnasally into the pharynx by a speech pathologist specializing in dysphagia management. FEES will be treated as a placebo comparator.

SUMMARY:
The purpose of this study is to determine if the Yale Swallow Protocol is an effective screen for aspiration in recently extubated patients.

DETAILED DESCRIPTION:
Dysphagia is prevalent in recently extubated patients with estimates ranging from 29-84% of recently extubated patients having some form of dysphagia with elevated risk for silent aspiration.One challenge providers face when managing post extubation dysphagia (PED) is that there are no best practice guidelines on how to evaluate for PED, specifically how to evaluate for silent aspiration (aspiration without cough response).

One method that has been suggested is the Yale Swallow Protocol (YSP), a pass/fail screen for aspiration consisting of a three ounce water challenge as well as a brief cognitive screen and oral motor exam. The assumption of the YSP is that silent aspiration (aspiration without a cough response) is volume dependent. This is based on a study of over 4000 patients that underwent both a FEES (5mL puree and 5mL liquid boluses) and a 3oz water challenge. Results from previous literature indicated that the 3oz water swallow had a high sensitivity for detecting aspiration (98%). This was again studied with a double blind research design with 25 patients, comparing results of the 3oz water challenge with results of videofluoroscopic swallow study. This showed 100% sensitivity for detecting aspiration, 64% specificity, 78% positive predictive value, and 100% negative predictive value. However, no published study has evaluated the YSP in recently extubated patients and so it is unclear if the high sensitivity and specificity would be retained. Investigators aim to determine the sensitivity and specificity of the Yale Swallow Protocol in identifying aspiration in recently extubated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Intubation greater than 24 hours
2. Age 18 and older
3. All races
4. Males and females
5. English speaking
6. Swallow consult ordered by the team within 48 hours of extubation

Exclusion Criteria:

1. Known history of oropharyngeal dysphagia
2. Contraindication for FEES due to facial fractures, nothing by mouth (NPO) status for other procedures, elevated bleeding risk, reduced level of alertness, or significant agitation.
3. Allergy to dairy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients recently extubated that are consulted for swallowing assessment by their treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Determine the sensitivity of the Yale Swallow Protocol (YSP) through aspiration identification in recently extubated patients. | Assessing the sensitivity of YSP within 2 study visit, within 2 hours. Data will be reported at study completion, an average of 1 year.
  Participants will receive FEES and YSP in a randomized order within a 2 hours of one another. Sensitivity estimates and analysis will be obtained through confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Stevie J Marvin, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States